CLINICAL TRIAL: NCT03351439
Title: Efficacy of Multimodal Analgesia Following Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Ryan Degen, Associate Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 110350
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hip Pain Chronic
Keywords: Hip Arthroscopy
MeSH Terms: interventions — zopiclone; Gabapentin; Celecoxib; oxycodone-acetaminophen; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Oxycodone-acetaminophen 5 mg/325 mg, 1-2 tabs every 6 hours as needed for 60 tabs Naprosyn 500 mg twice daily x 3 weeks
  Interventions: Drug: Percocet; Drug: Naprosyn
- Group 2 (Experimental): Oxycodone-acetaminophen 5 mg/325 mg, 1-2 tabs every 6 hours as needed for 60 tabs Naprosyn 500 mg twice daily for 3 weeks Zopiclone 7.5 mg nightly for 7 days
  Interventions: Drug: Zopiclone; Drug: Percocet; Drug: Naprosyn
- Group 3 (Experimental): Oxycodone-acetaminophen 5 mg/325 mg, 1-2 tabs every 6 hours as needed for 60 tabs Naprosyn 500 mg twice daily for 3 weeks Gabapentin 600 mg pre-operatively for one dose and 600 mg post-operatively for one dose
  Interventions: Drug: Gabapentin; Drug: Percocet; Drug: Naprosyn
- Group 4 (Experimental): Oxycodone-acetaminophen 5 mg/325 mg, 1-2 tabs every 6 hours as needed for 60 tabs Naprosyn 500 mg twice daily for 3 weeks Celebrex 400 mg pre-operatively for one dose
  Interventions: Drug: Celebrex; Drug: Percocet; Drug: Naprosyn

INTERVENTIONS:
Drug: Zopiclone — Group 2 - Zopiclone 7.5 mg orally, nightly for 7 days
  Arms: Group 2
Drug: Gabapentin — Group 3 - Gabapentin 600 mg orally, 1 hour pre-operatively and 600 mg orally, 8 hours post-operatively
  Arms: Group 3
Drug: Celebrex — Group 4 - Celebrex 400 mg PO, 1 hour pre-operatively
  Arms: Group 4
Drug: Percocet — Standard of Care
Drug: Naprosyn — Standard of Care

SUMMARY:
The purpose of the full study is to determine whether multimodal analgesia for hip arthroscopy will reduce post-operative pain scores, narcotic consumption and hospital length-of-stay. To do this, the investigators will compare the standard of care (SOC), with routine pain management with a post-operative opioid prescription, to three different groups with multi-modal analgesia (SOC+peri-operative celecoxib, SOC+peri-operative gabapentin, and SOC+post-operative zopiclone).

The investigators hypothesize that administration of multi-modal analgesia in all three treatment groups will result in improved post-operative pain control, reduced post-operative narcotic consumption and an overall reduction in post-operative length-of-stay compared to the group receiving treatment as per the standard of care. However, prior to undertaking a large multi-centre study, the investigators need to determine whether the study is feasible from data obtained with this pilot study.

DETAILED DESCRIPTION:
This pilot study will be a randomized controlled trial, where the surgical team, data collector, and patient will be blinded to the treatment received. The investigators will include any patient between the ages of 18 and 60 years undergoing hip arthroscopy by one of three fellowship-trained hip arthroscopists. The investigators will exclude patients with any radiographic signs of osteoarthritis (Tönnis grade 2 or higher), an American Society of Anesthesiologists (ASA) classification of 3 or higher, allergies to sulfa-based drugs, adverse reactions to any of the potential study medications, or a history of chronic pain or substance abuse.

Patients will be randomized in a 1:1:1:1 ratio into one of four groups:

1. Group 1 - Standard of Care (SOC): Opioid medication (Oxycodone-acetaminophen 5 mg/325 mg, 1-2 tabs every 6 hours as needed), Heterotopic ossification prophylaxis - Naprosyn 500 mg twice daily x 3 weeks);
2. Group 2 - SOC + Post-operative sleeping aid (Zopiclone 7.5 mg nightly x 7 days);
3. Group 3 - SOC + Pre-operative and Post-operative Gabapentin (600 mg orally, 1 hour pre-operatively; 600 mg 8 hours post-operatively);
4. Group 4 - SOC + Pre-medicate with Celebrex (400 mg orally, 1 hour pre-operatively)

A member of the research team will ensure that the surgeons, data collectors, and patients remain blinded to the treatment group and by performing all randomization and medication administration. For those patients randomized to the celebrex or gabapentin groups, a dose of each respective medication will be administered 1 hour before arthroscopic surgery. To maintain blinding, patients in the SOC group and zopiclone groups will receive a lactose-based placebo at the same time. Post-operatively, patients randomized to the zopiclone group will receive a prescription to be taken at night. Patients in the other three groups will receive lactose-based placebo pills for the same duration, again to maintain blinding.

All patients will receive similar treatment for their hip arthroscopy. All surgeries will be performed in the supine position utilizing a hip distraction system (Smith and Nephew, Andover MA). The procedure will be performed with use of a general anesthetic without regional anesthesia. Pathology will be identified and treated at the discretion of the primary surgeon. Patients will receive a standardized anesthetic regimen intra-operatively. Portal sites will be injected with a total of 20cc of bupivacaine. Following the procedure, all patients will be managed with a standardized post-operative analgesic regimen and subsequently discharged with a prescription for oral analgesics and prophylaxis against heterotopic ossification. Patients will be instructed to retain and return any unused narcotics at subsequent follow-up at the 2-week post-operative visit. Patients will be encouraged to request additional prescriptions through their surgeons' office for tracking, although a chart review will be performed to evaluate for any additional emergency department visits post-operatively.

The investigators will collect demographic information, including age and sex, and intra-operative data as to the surgical procedures performed including potential confounders like the duration of traction time, and dose of intraoperative narcotics. The investigators will measure pain preoperatively using a pain visual analog scale (VAS). Postoperatively, patients will again be evaluated for pain with using the same VAS at 1 hour, 2 hours, 6 hours, 24 hours, daily for 7 days and every other day for 6 weeks. Post-operatively, in hospital complications including nausea/vomiting/urinary retention will be recorded. Patient satisfaction will also be evaluated at 24 hours, 48 hours, daily for 7 days and every other day for 6 weeks. The total quantity of narcotics consumed will be calculated after accounting for unused medications returned post-operatively and additional prescription requests. Lastly, the hospital length-of-stay and associated costs will be calculated form the patients hospital records. Patients will also be administered a questionnaire on cost-reporting to evaluate for any costs due to visits to any emergency room, other physician, additional visits to rehabilitation or pain specialists, additional medications including over-the-counter medications obtained by the patient or those prescribed by another physician on a weekly basis for 6 weeks.

The investigators will consecutively approach all patients undergoing a hip arthroscopy until 100 patients are eligible and give their consent to participate (approximately one year from study commencement). This number of patients will provide a sufficient sample size to accurately estimate the proportion of eligible patients who will give their consent (the study will be sufficiently powered to provide the estimate with a 95% confidence interval around the estimate where half the width of the confidence interval [CI] is no greater than 0.05).

ELIGIBILITY:
Inclusion Criteria:

* any patient between the ages of 18 and 60 years undergoing hip arthroscopy by one of three fellowship-trained hip arthroscopists

Exclusion Criteria:

* radiographic signs of osteoarthritis (Tönnis grade 2 or higher), an American Society of Anesthesiologists (ASA) classification of 3 or higher,
* allergy to sulfa-based drugs,
* adverse reactions to any of the potential study medications, or a
* history of chronic pain, substance abuse or
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score | Baseline, 1, 2, 6, 24hr post-op, daily for 1 week, every other day for 6 weeks
  Visual Analog Scale 0-100 to determine daily hip pain; 0=extreme pain, 100=no pain

SECONDARY OUTCOMES:
Change in Patient Satisfaction | Daily for 1 week, every other day for 6 weeks
  Visual Analog Scale 0-100 to determine satisfaction with pain control; 0=extremely dissatisfied; 100=extremely satisfied
Change in Length of Stay | 24 hrs
  Records the length of stay in hospital post-operative
Change in Post-operative Complication Rates | 24 hours
  Records any post-op complications
Change in Post-operative Narcotic Consumption | 2 weeks
  Diary to record pain medication consumption
Cost Diary | Weekly for 6 weeks
  Patient reported diary to record hospital and personal expenses

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Degen, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada